CLINICAL TRIAL: NCT07362589
Title: The Effect of Pain Education Given to Patients Before Total Knee and Hip Replacement Surgery on Anxiety, Pain and Analgesic Use: A Randomized Controlled Study
Brief Title: Effect of Preoperative Pain Education on Anxiety, Pain, and Analgesic Use in Total Knee and Hip Replacement Patients
Acronym: Pain-Anxiety
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Ceren Ustun, Hemşire Ceren Üstün, Yeditepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: E.83321821-805.02.03-472
Record Dates: First submitted 2025-09-23; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Pain Management; Arthroplasty; Knee Replacement; Hip Replacement
Keywords: Postoperative Pain; Nursing; Patient Education
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Pain Education
  Interventions: Other: Pain education
- Control Group (No Intervention): No education no video

INTERVENTIONS:
Other: Pain education — education booklet and video
  Arms: Experimental Group

SUMMARY:
This randomized controlled trial evaluates whether a standardized preoperative pain education session delivered by a nurse reduces postoperative pain intensity and surgical anxiety among adult elective orthopedic surgery patients compared with usual care.

Primary outcome is postoperative pain at 24 hours. Secondary outcomes include anxiety, analgesic consumption, patient satisfaction, and length of stay

DETAILED DESCRIPTION:
Adult patients scheduled for elective orthopedic surgery will be randomized (1:1) to receive either (a) a structured 20-30-minute preoperative pain education session plus booklet and video, or (b) usual care alone. Pain intensity measured with NRS at 1, 6,12, 24, 48h postop; analgesics recorded Day 0, 1, 2; preop anxiety measured with Surgical Anxiety Scale in both groups. Intention-to-treat analysis.

ELIGIBILITY:
Inclusion criteria:

* Being 18 years of age or older,
* Providing voluntary informed consent to participate in the study,
* Scheduled to undergo elective knee or hip joint replacement (arthroplasty) surgery,
* Having no communication barriers,
* Having no history of alcohol or substance dependence,
* Having no concurrent diagnosis of malignant disease and not receiving cancer treatment,
* Not using opioid medications regularly in the preoperative period,
* Having an ASA score of III or below,
* Having no cognitive impairment that would affect the ability to comprehend the provided education,
* Having no diagnosed neurological or psychiatric disorder and not using medications related to such conditions.

Exclusion criteria:

- Patients who do not meet the specified inclusion criteria will not be included in the study.

Elimination criteria:

* Indication for postoperative intensive care,
* Development of major complications after surgery, such as massive bleeding or pulmonary embolism,
* Requesting to withdraw from the study at any stage,
* Use of a patient-controlled analgesia device postoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Is there a difference in postoperative pain levels between the intervention group, which received preoperative pain education, and the control group, which did not receive preoperative pain education?" | Pain assessment was evaluated at 1, 6, 12, 24, and 48 hours postoperatively.
  The intervention group received a preoperative pain education booklet and watched a pain education video, while the control group did not receive any educational intervention. Both groups were asked to rate their pain on the Numerical Rating Scale (NRS) from 0 to 10 at 1, 6, 12, 24, and 48 hours postoperatively, where 0 indicated no pain (a good score) and 10 indicated the worst possible pain (a poor score). Since pain is subjective, the patients' self-reported scores were recorded as provided. The differences between the two groups were subsequently analyzed.
Does preoperative pain education reduce preoperative anxiety? | Baseline (preoperatively, before surgery) and postoperatively at 1 hour, 6 hours, 12 hours, 24 hours, and 48 hours after surgery.
  This study aims to investigate whether there is a significant difference in preoperative anxiety levels between patients who received preoperative pain education (intervention group) and those who did not (control group). The Surgical Anxiety Questionnaire - (SAQ) was used to assess patients anxiety.
  In this 17-item scale, the individual is asked to rate how anxious or worried they are for each item on a five-point likert type scale:"Not at all", "A little bit" ''Moderately'' ''Very'' and ''Extremely''. The answers given to each item are scored between 0-4. There is no cut-off value, and as the score increases, the individual anxiety is interpreted as higher. Cronbachs alpha coefficient was reported to be 0.91 in the original version of the scale. The Turkish version of the surgical anxiety questionnaire consisted of a 3-factor structure, and the Cronbach alpha value was 0.93. As a result, the Turkish form of the scale contains 15 items.

CONTACTS AND LOCATIONS:
Overall Officials: İNCİ KIRTIL, Assist.Prof, Study Director — Yeditepe Üniversitesi
Locations (1):
- Yeditepe Üniversitesi Hastanesi, Istanbul, Kayişdaği, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Decision not reached
Supporting Information: Study Protocol, SAP, ICF

DOCUMENTS (1):
  • Informed Consent Form (2025-09-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT07362589/ICF_000.pdf